CLINICAL TRIAL: NCT04441073
Title: Lignocaine Nebulization for Attenuation of Intubation Stress Response in Patients With Severe Pre-eclampsia: a Prospective Double-blinded Placebo-controlled Trial
Brief Title: Lignocaine Nebulization for Attenuation of Intubation Stress Response
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, FATMA NABIL AHMED MOHAMED, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Lignocaine nebulization stress
Record Dates: First submitted 2020-06-05; First posted 2020-06-22 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Pressor Response
Keywords: pressor response; pre-eclampsia; Lignocaine
MeSH Terms: conditions — Pre-Eclampsia | interventions — Lidocaine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lignocaine (Experimental): preoperative nebulization of lignocaine
  Interventions: Drug: Lignocaine
- Placebo (Placebo Comparator): preoperative nebulization of normal saline (Nacl 0.9%) as a placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lignocaine — preoperative nebulization of lignocaine
  Arms: Lignocaine
Drug: Placebo — preoperative nebulization of normal saline (Nacl 0.9%) as a placebo
  Other Names: Normal saline (Nacl 0.9%)
  Arms: Placebo

SUMMARY:
To study the effect of lignocaine nebulization on attenuation of the pressor response during induction and emergence of anesthesia in patients with severe pre-eclampsia

DETAILED DESCRIPTION:
The pressor response to laryngoscopy and tracheal intubation is a very important issue in hypertensive pregnant patients that can lead to increased maternal intracranial pressure, cerebral haemorrhage, and cardiac failure with pulmonary oedema and may result in maternal mortality. The catecholamine release associated with laryngoscopy and intubation also causes uteroplacental vasoconstriction and adversely affect the neonate well-being.

Therefore, the precise control of stress is necessary during general anesthesia in pre-eclamptic patients.Various drugs are used to suppress the pressor response including opioids, lidocaine, along with α and β adrenergic blockers.

in this study the investigators will evaluate the effect of lignocaine nebulization on attenuation of the pressor response.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist (ASA) II , III with severe pre-eclampsia
* Scheduled for caesarean deliveries under general anesthesia

Exclusion Criteria:

* severe obesity (BMI ≥ 40 )
* Cardiac patients
* History of diabetes
* Renal dysfunction (Elevated creatinine ≥ 2 mg\dl)
* Hepatic dysfunction (Elevated hepatic enzymes three times above normal value)
* Known fetal anomalies

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-02-24 (Actual); Primary Completion 2022-02-23 (Estimated); Study Completion 2022-02-23 (Estimated)

PRIMARY OUTCOMES:
Systolic, diastolic, mean arterial blood pressure | Preoperative-Intraoperative
Heart rate | Preoperative-Intraoperative
Peripheral oxygen saturation | Preoperative-Intraoperative
Cough score during emergence | Up to one hour after extubation
  Grade of coughing (grade 0: no cough; grade 1: single cough with mild severity; grade 2: cough lasting less than 5 seconds with moderate severity; grade 3: more than 5 seconds of persistent cough)

SECONDARY OUTCOMES:
APGAR score | One, 5 and 10 minutes after delivery of the fetus
  APGAR stands for "Appearance, Pulse, Grimace, Activity, and Respiration."
  In the test, five things are used to check a baby's health. Each is scored on a scale of 0 to 2, with 2 being the best score
Sore throat and hoarseness of voice | Postoperative (one, 6 and 24 hours)
  The incidences and severities of postoperative sore throat and hoarseness of voice will be measured using direct questions

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided